CLINICAL TRIAL: NCT00425165
Title: A Randomized, Double-Blind, Two Way Crossover Evaluation of the Effects of a Single Dose of Denufosol Tetrasodium (INS37217) Inhalation Solution Versus Placebo (0.9% Sodium Chloride Solution) on Mucociliary Clearance in Patients With Mild to Moderate Cystic Fibrosis Lung Disease
Brief Title: Study of Denufosol Inhalation Solution in Patients With Mild to Moderate Cystic Fibrosis Lung Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-111
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Inhalation Solution — Denufosol 60 mg is administered as an inhalation solution one time during the study.

SUMMARY:
The purpose of this trial is to evaluate the effects of a single dose of denufosol versus placebo on mucociliary clearance in patients with mild to moderate CF lung disease

ELIGIBILITY:
Inclusion Criteria:

* have confirmed diagnosis of cystic fibrosis
* have FEV1 of greater than or equal to 60% of predicted normal for age, gender, and height
* be able to reproducibly perform spirometry maneuvers
* be clinically stable for at least 4 weeks prior to screening

Exclusion Criteria:

* have abnormal renal or liver function
* have chest x-ray at screening with abnormalities suggesting clinically significant active pulmonary disease
* have had a lung transplant

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in mucociliary clearance from baseline | 30, 60, and 90 minutes post aerosol inhalation